CLINICAL TRIAL: NCT00397384
Title: A Phase I Clinical and Biological Evaluation of Combined EGFR Blockade With Erlotinib and Cetuximab in Patients With Advanced Cancer
Brief Title: Erlotinib Hydrochloride and Cetuximab in Treating Patients With Advanced Gastrointestinal Cancer, Head and Neck Cancer, Non-Small Cell Lung Cancer, or Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00107; NCI-2009-00107 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000511880; GI 0622 (Other: Vanderbilt-Ingram Cancer Center); 6980 (Other: CTEP); P30CA068485 (NIH)
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2014-02

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Advanced Adult Primary Liver Cancer; Carcinoma of the Appendix; Gastrointestinal Stromal Tumor; Metastatic Gastrointestinal Carcinoid Tumor; Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Adult Primary Liver Cancer; Recurrent Anal Cancer; Recurrent Basal Cell Carcinoma of the Lip; Recurrent Colon Cancer; Recurrent Esophageal Cancer; Recurrent Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Recurrent Extrahepatic Bile Duct Cancer; Recurrent Gallbladder Cancer; Recurrent Gastric Cancer; Recurrent Gastrointestinal Carcinoid Tumor; Recurrent Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Recurrent Lymphoepithelioma of the Nasopharynx; Recurrent Lymphoepithelioma of the Oropharynx; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Non-small Cell Lung Cancer; Recurrent Pancreatic Cancer; Recurrent Rectal Cancer; Recurrent Salivary Gland Cancer; Recurrent Small Intestine Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Small Intestine Adenocarcinoma; Small Intestine Leiomyosarcoma; Small Intestine Lymphoma; Stage IV Adenoid Cystic Carcinoma of the Oral Cavity; Stage IV Anal Cancer; Stage IV Basal Cell Carcinoma of the Lip; Stage IV Colon Cancer; Stage IV Esophageal Cancer; Stage IV Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage IV Gastric Cancer; Stage IV Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage IV Lymphoepithelioma of the Nasopharynx; Stage IV Lymphoepithelioma of the Oropharynx; Stage IV Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage IV Mucoepidermoid Carcinoma of the Oral Cavity; Stage IV Non-small Cell Lung Cancer; Stage IV Pancreatic Cancer; Stage IV Rectal Cancer; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity; Tongue Cancer; Unresectable Extrahepatic Bile Duct Cancer; Unresectable Gallbladder Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Appendiceal Neoplasms; Gastrointestinal Stromal Tumors; Carcinoma, Hepatocellular; Anus Neoplasms; Esophageal Neoplasms; Esthesioneuroblastoma, Olfactory; Bile Duct Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Cetuximab; Erlotinib Hydrochloride

ARMS (1):
- Treatment (cetuximab and erlotinib hydrochloride) (Experimental): Patients receive cetuximab IV over 1-2 hours on days 1, 8, and 15 and erlotinib hydrochloride PO QD on days 8-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cetuximab; Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of erlotinib hydrochloride when given together with cetuximab and to see how well they work in treating patients with advanced gastrointestinal cancer, head and neck cancer, non-small cell lung cancer, or colorectal cancer. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Erlotinib hydrochloride and cetuximab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving erlotinib hydrochloride together with cetuximab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the maximum tolerated dose (MTD). II. To identify the recommended dose (RD) for phase II of erlotinib (erlotinib hydrochloride) in combination with cetuximab in patients (pts) with incurable gastrointestinal, head and neck, or non-small cell lung cancers that are Kirsten rat sarcoma viral oncogene homolog (KRAS) wild type.

SECONDARY OBJECTIVES:

I. To identify dose-limiting toxicities (DLT). II. To perform skin and tumor biopsies to analyze molecular inhibition of the epidermal growth factor receptor (EGFR) signaling pathway, defined as a >= 75% inhibition of phosphorylation of the epidermal growth factor (EGF) receptor or of its downstream effectors tumor protein (p)44/42 mitogen-activated protein kinase (MAPK) or protein kinase B (Akt) or as a >= 25% decrease of marker of proliferation Ki-67 (Ki67) from baseline in either skin or tumor tissue in the majority of patients.

III. To identify the optimal biological dose (OBD). IV. To describe any antitumor effect observed.

OUTLINE: This is a phase I, dose-escalation study of erlotinib hydrochloride.

Patients receive cetuximab intravenously (IV) over 1-2 hours on days 1, 8, and 15 and erlotinib hydrochloride orally (PO) once daily (QD) on days 8-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed incurable gastrointestinal tract, head and neck, or non-small cell lung cancers that are KRAS wild type; if KRAS mutational status cannot be determined on archived tumor tissue from the patient, a needle or excisional biopsy of a malignant site may be performed prior to enrollment; mutational status may be determined either by polymerase chain reaction (PCR) assay (e.g., DxS KRAS mutation kit) or by direct sequencing of KRAS exon 2, codons 12 and 13; the result must detect no mutations at these sites
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits or creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of erlotinib will be determined following review of their case by the principal investigator; although concomitant use of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducers is not prohibited in this study, identification of MTD and DLT may be affected by their use; concomitant use of any of these drugs will be noted in the case report forms and will be taken into account in determining MTD and DLT of this therapy; efforts should be made to switch patients with a history of brain metastases who are taking enzyme-inducing anticonvulsant agents to other medications
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Other prior malignancies are allowed provided prior therapy has been discontinued and there is no evidence of disease (NED)
* Patients must be able to take and retain oral medications
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with a history of brain metastases are eligible provided that the metastases have been surgically resected and/or are radiographically and clinically stable for 2 months following the completion of radiation therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cetuximab
* Prior treatment with EGFR-targeting therapies
* Major surgery or significant traumatic injury occurring within 21 days prior to treatment
* Abnormalities of the cornea based on history (e.g., dry eye syndrome, Sjogren's syndrome), congenital abnormality (e.g., Fuch's dystrophy), abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal-Rose), and/or an abnormal corneal sensitivity test (Schirmer test or similar tear production test)
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with erlotinib or cetuximab
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Incidence of DLT, defined as recurring grade 2 or greater non-hematological or grade 3 or greater hematological toxicities or skin rash graded using Common Terminology Criteria for Adverse Events version 3.0 (CTCAE-v3) | 21 days
MTD defined as the dose level at which fewer than 2 out of 6 patients experience DLT graded using CTCAE-v3 | 21 days

SECONDARY OUTCOMES:
Change in molecular inhibition of the EGFR signaling pathway | Baseline to up to 4 weeks
  These data will be descriptive in nature, with no hypothesis testing. Summary statistics including numbers of subjects that met response criteria, and mean, median and standard deviation in the percent staining, all by dose level.
OBD defined as the dose at which either a >= 75% inhibition of phosphorylation of the EGF receptor or of its downstream effectors p44/42 MAPK or Akt is observed, or Ki67 is decreased by >= 25% | Up to 4 weeks
  These data will be descriptive in nature, with no hypothesis testing. Summary statistics including numbers of subjects that met response criteria, and mean, median and standard deviation in the percent staining, all by dose level.
Antitumor effect observed | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laura Goff, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States